CLINICAL TRIAL: NCT04892316
Title: Using Machine Learning to Adapt Visual Aids for Patients With Low Vision
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: SFLV-2020
Record Dates: First submitted 2021-05-17; First posted 2021-05-19 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Ophthalmology; Artificial Intelligence; Low Vision Aids
Keywords: Artificial Intelligence; Low Vision
MeSH Terms: conditions — Vision, Low | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Junior doctor group: Patients receive assisting devices fitting services from junior doctors
  Interventions: Diagnostic Test: Diagnostic test
- Senior doctor group: Patients receive assisting devices fitting services from senior doctors
  Interventions: Diagnostic Test: Diagnostic test
- Algorithm assisted group: Patients receive assisting devices fitting services from junior doctors assisted by the machine learning model
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — The training dataset was used to train the model, which was validated and tested by the other two datasets.

SUMMARY:
According to the WHO's definition of visual impairment, as of 2018, there were approximately 1.3 billion people with visual impairment in the world, and only 10% of countries can provide assisting services for the rehabilitation of visual impairment. Although China is one of the countries that can provide rehabilitation services for patients with visual impairment, due to restrictions on the number of professionals in various regions, uneven diagnosis and treatment, and regional differences in economic conditions, not all visually impaired patients can get the rehabilitation of assisting device fitting.

Traditional statistical methods were not enough to solve the problem of intelligent fitting of assisting devices. At present, there are almost no intelligent fitting models of assisting devices in the world. Therefore, in order to allow more low-vision patients to receive accurate and rapid rehabilitation services, we conducted a cross-sectional study on the assisting devices fitting for low-vision patients in Fujian Province, China in the past five years, and at the same time constructed a machine learning model to intelligently predict the adaptation result of the basic assisting devices for low vision patients.

ELIGIBILITY:
Inclusion Criteria:

* Low vision
* Aged 3 to 105

Exclusion Criteria:

* Severe systemic disease
* Failure to sign informed consent or unwilling to participate

Ages: 3 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Visually disabled patients were referred by the Town Disability Federation in Fujian Province and Guangdong Province
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-07-27 (Estimated); Study Completion 2021-12-27 (Estimated)

PRIMARY OUTCOMES:
Accuracy of fitting results for assisting devices | baseline
  The investigator will calculate the accuracy of fitting results for assisting devices in different group according to the ground truth.

SECONDARY OUTCOMES:
Time cost for fitting assisting devices | baseline
  The investigator will calculate time cost for fitting assisting devices in different group.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affilliated Hospital of Fujian Medical University, Quanzhou, Fujian, China